CLINICAL TRIAL: NCT02446652
Title: Phase III Clinical Trial: "Evaluation of the Combination of TRANSKRIP ® Plus Carboplatin and Paclitaxel as First Line Chemotherapy on Survival of Patients With Recurrent - Persistent Cervical Cancer
Brief Title: Evaluation of TRANSKRIP ® Plus Chemotherapy in Recurrent-Persistent Cervical Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a lack of sufficient resources, the opening was not carried out.
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Psicofarma, S.A. De C.V. (Industry)
Responsible Party: Principal Investigator, Lucely Cetina Pérez, MD. MSc., National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (014/037/ICI)(CEI/941/14)
Record Dates: First submitted 2015-04-20; First posted 2015-05-18 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
Keywords: Advanced cervical cancer; Epigenetic therapy; Randomized phase III
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Hydralazine; Magnesium; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydralazine/Magnesium valproate + QT (Experimental): This group will receive TRANSKRIP® (Hydralazine/Magnesium valproate) + Carboplatin plus Paclitaxel
  Interventions: Drug: Hydralazine/Magnesium; Drug: Carboplatin; Drug: Paclitaxel
- placebo + QT (Placebo Comparator): This group will receive placebo + Carboplatin plus Paclitaxel
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Hydralazine/Magnesium — (Hydralazine: 1 oral tablet every 24 hours, 182 mg for rapid acetylators, and 83 mg for low acetylators and Magnesium valproate: orally 30 mg/K weight every 8 hours) starting 1 week prior the first day of the QT
  Other Names: TRANSKRIP ®
  Arms: Hydralazine/Magnesium valproate + QT
Drug: Placebo — Placebo (orally) starting 1 week before the first day of the QT
  Arms: placebo + QT
Drug: Carboplatin — 5 AUC 1 hour/day 1 for every 21 days for 6 cycles
  Other Names: CBP
Drug: Paclitaxel — 175mg/m2/SC 3hour/day 1 for every 21 days for 6 cycles.
  Other Names: PXL

SUMMARY:
The purpose of this study is to determine the efficacy and safety the combination of TRANSKRIP ® vs placebo plus Carboplatin/Paclitaxel as first line treatment in patients with recurrent-persistent cervical cancer.

DETAILED DESCRIPTION:
HYPOTHESIS: It is estimated that adding TRANSKRIP ® to the chemotherapy an increase will occur in the survival of at least 3.6 months superior compared to the patients receiving only QT (17.9 months for TRANSKRIP plus QT and 14.3 months for QT, i.e. a 20% of difference).

Sample size: Data from GOG (Gynecologic Oncology Group) 240 study was used to define it where at 36 months the survival rate was 39.5% for the control group. Losses of 20%, 95% α, 80% β, among groups of 1 ratio and a better 20% survival in the experimental group were considered. From the above, 230 are included which will be in blocks of 10.

Study overview: In patients who meet the inclusion criteria an informed consent oral and written will be granted, once accepted screening test will be made to determine exclusion criteria (CAT, laboratories). If they meet all criteria, patients will be assigned to the following treatment groups:

Group A (115 patients): TRANSKRIP® (Hydralazine: 1 oral tablet every 24 hours, 182 mg for rapid acetylators, and 83 mg for low acetylators and Magnesium valproate: orally 30 mg/K weight every 8 hours) starting 1 week prior the first day of the QT Carboplatin based (5 area under curve (AUC) 1hour/day 1) plus Paclitaxel (175 175mg/m2/body surface (BS) 3hour/day 1) for every 21 days for 6 cycles.

Group B (115 patients): Placebo (orally) starting 1 week before the first day of the QT Carboplatin based (5 AUC 1hour/day 1) plus Paclitaxel (175 175mg/m2/BS 3hour/day 1) for every 21 days for 6 cycles.

Patients included in the study will be conducted to determine their acetylator genotype by polymerase chain reaction (PCR) sequencing N-acetyltransferase 2 (NAT2) gene, and blood samples will be sent to the central laboratory CIDAT S.A de C.V. Those with slow acetylation result will receive 83 mg/day of Hydralazine plus 30 mg/Kg/day of magnesium Valproate, patients with fast acetylation result will receive 182 mg/day of Hydralazine plus 30 mg/Kg/day of magnesium Valproate.

Assigning patients: Randomization will be automatically generated in a computer and with the randomization program; the list will be generated by the Contract Research Organization (CRO) hired for this study. The flasks will be labeled by the Alpharma Manufacturing Department, from the random list that identifies the treatment that every patient receives.

Dose adjustments: All patients should have, previous to the chemotherapy administration, an absolute neutrophil count >1500/µL and platelets greater than 100,000/µL. If they have smaller numbers, treatment will be delayed during 1-2 weeks, until achieving these levels. There won't be dose adjustment of the chemotherapy. The chemotherapy dosage should not exceed the initial dose calculation, unless the patient has a weight change greater than 10% requiring the new dose calculation. A patient which cannot take the drug during 6 weeks since the last treatment should be discontinued from the study. In case of renal toxicity grade 3-4, the dosage of carboplatin will be decreased to 50%.

Dose reduction of magnesium Valproate: If a patient shows somnolence grade 3 and/or ataxia grade 3 magnesium valproate will be suspended for 3 days or until the toxicity is at least grade 2 and will restart to 20 mg/Kg. If after 7 days somnolence grade 3 is not presented it will be increased to 30 mg/Kg and will continue with this dose until the end of the study. If toxicity grade 3 is resubmitted the patient will continue with 20 mg/Kg until the end of the study.

Dose reduction of hydralazine: If a patient shows hypotension grade 3, hydralazine will be suspended for 3 days or until the toxicity is at least grade 2 and will restart to 50% of the dose. If after 7 days hypotension grade 3 is not presented it will increase to 100% of the dose and will continue with this dose until the end of the study.

Procedures No more than 14 days before the initiation of study drug, the state of the disease form every patient will be evaluated with the following procedures: Medical history and physical examination,Evaluation of the performance status (ECOG scale), complete blood count (CBC), Blood chemistry, Liver Function test (LFT), Electrolytes, antinuclear antibodies, Measurement of palpable or visible lesions, as well as those determined by imaging studies by computed tomography of the abdomen, thorax and pelvis, Quality of life questionnaires will be applied to know their basal state.

At the beginning of each cycle: Medical history and physical examination, Evaluation of the performance status (ECOG scale), CBC, Blood chemistry, LFT, Electrolytes, antinuclear antibodies, Hydralazine levels and valproic acid in blood (every 2 cycles), Toxicity evaluation with the established criteria by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE V.3.0).

At the end of 3 and 6 cycles: Medical history and physical examination, Evaluation of the performance status (ECOG scale), CBC, Blood chemistry, LFT, Electrolytes, antinuclear antibodies, Measurement of palpable or visible lesions, as well as those determined by imaging studies by computed tomography, Quality of life questionnaires (QLQ) Cx-30 and C-24 will be applied.

Follow up visits post-treatment will be every 3 months the first 2 years, every 4 months the third year, every 6 months the fourth year and later annually or until progression. During this period Clinical History and physical examination, assessment of performance status, weight and tumor lesion measurements by physical examination or by imaging studies will be obtained. CBC, Blood chemistry, LFT, electrolytes and antinuclear antibodies. Relapse, progression or recurrence date. Quality of life will be evaluated every 6 months during follow to complete 2 years of starting the patient in the study.

Patients will participate in this study during the period prior to treatment and during the QT (Carboplatin plus paclitaxel) administration, or until the experimental treatment with TRANSKRIP® vs Placebo is suspended. Patients may withdraw from the study by progression of the disease, intolerable toxicity, withdrawal of consent by the patient or investigator decision to suspend the participation of the patient in the study. In case of suspending the treatment, patient will continue monitoring or under non-protocol treatment by the treatment service.

Efficacy criteria. The measuring tumor (s) is defined as: Dimensionally measurable: The minimum size of the lesion to be considerable measurable s 10 mm if the cuts from the scanner are of at most 5mm and 20mm with higher cuts of 5mm. A maximum of 5 blank lesions by organ and/or 10 total lesions will be identified. The sum of the maximum diameters from each of the lesions will be considered as the basal measure from the sum of the maximum diameters and this number will be used to categorize the answer. Unidimensionally measurable disease, lesions in previously irradiated fields, ascites, pleural effusions, bone, blastic or mixed metastases or abdominal masses that can be palpated but not measured shall not be considered measurable. To determine the disease status during the study will be evaluated by RECIST criteria.

Clinical Adverse Events: Initially, the staff study site will interrogate each patient and will write the occurrence and nature of the condition (s) of presentation and any preexistent condition (s). During the study, the staff will interrogate the patient and will write any change in the preexistent condition (s) and/or the occurrence and nature of any adverse event. All the adverse events should be reported to the regulatory agency and to the appropriated pharmaceutical companies according to the local regulations.

The staff study site should report to the local regulatory body (COFEPRIS and to the respective committees of the National Cancer Institute), any severe adverse event possibly related to the study drugs including: death, initial or prolonged hospitalization, laying in life threatening, severe or permanent disability or congenital anomaly.

Patient substitution: It is considered replaceable, any patient that has been randomized, but for some reason it has not receive any doses of Transkrip vs placebo, to not affect the trust and power of the sample.

Statistical analysis: All patients who receive the first cycle of chemotherapy study will be evaluated for safety.

All patients who meet histological diagnosis of cancer, presence of dimensionally measurable disease and evaluation with computed axial tomography (CAT) and/or Magnetic Resonance Imaging (MRI) after the third cycle will be evaluated for efficacy.

All confidence intervals will be built with a level of significance of α = 0.05 (Confidence level of 95%). One interim analysis is expected and one final analysis, the first one after included the first 115 patients and upon completion the QT, final analysis is expected at 19 months that the last patient has been included. Intention analysis to treatment to all patients included and by protocol to those who meet the criteria for analysis will be carried out.

Processing and analysis of the data base will be made with the Statistical Package for the Social Sciences (IBM SPSS) version 19.0 ® for Microsoft. The demographic, clinical, of treatment and disease characteristics, will be analyzed, through descriptive statistics: measures of central and dispersion tendency: range, measure, median, mode, standard deviation, proportions and ratios.

Global Survival. It is considered as an initial event the subject inclusion in the study and final event of death. Survival times will be estimated by the no parametric estimator of Kaplan-Meier. Variances and confidence intervals for those will be estimated. Survival curves will be compared by logrank test, considering a bilateral test, and the significance level of 95%. Format Cox regression will be applied to evaluate the influence of control variables in the survival time. Also survival times will be calculated considering as an initial event the disease diagnose and progression.

Objective Response: for parameters for nominal and ordinal scale Chi square test or Fisher exact will be used. For quantitative variables or intervals T Student test will be used if homogeneity.

Toxicity: incidence of adverse effects will be estimated, as well as their frequency by severity, the laboratory values during treatment. Frequency of abnormal laboratory values will be estimated.

Quality of life: The linear transformation of the data was performed to obtain values on a scale of 0-100. In the case of missing data, the calculation of gross score in both the numerator and denominator, will be made taking into account only the items with response. Thus avoiding the values are affected by extremes. Baseline analysis between groups by obtaining mean and standard deviation or median and interquartile ranges, after analysis of data normality by Kolmogorov-Smirnov took place. The bivariate analysis was evaluated by student test for independent samples when the data is parametric or Mann Whitney test for nonparametric data. With an alpha of 0.05 two-tailed. Besides an intragroup longitudinal analysis will be performed to monitor changes in the quality of life through% change between the first and second assessment and bivariate analysis using paired t or Wilcoxon. With an alpha of 0.05 two-tailed.

Progression free survival: It is considered as an initial event the subject inclusion in the study and final event the progression of disease. Survival times will be estimated by the no parametric estimator of Kaplan-Meier. Variances and confidence intervals for those will be estimated. Survival curves will be compared by logrank test, considering a bilateral test, and the significance level of 95%. Format Cox regression will be applied to evaluate the influence of control variables in the survival time.

ELIGIBILITY:
Inclusion Criteria:

* Operating status ECOG: 0-2
* Negative pregnancy test or reproduction potential is zero, determined either by surgery, radiation or menopause, or mitigated with the use of some approved contraceptive method (IUD or hormonal contraceptive during the study and at least 3 months after the study).
* Patients with histological diagnosis of persistent/recurrent cervical cancer, local and/or systemic, with disease measurable by physical examination and TAC. REQUIRED confirmation by biopsy of the recurrence or, persistence only if: lesion is single, less than 2 cm and/or has no sharp edges.
* Chemo-radiotherapy to pelvis or pelvis plus extended fields (may have received concomitant chemotherapy as a radiosensitizer) provided it is within 90 days from the last application and the secondary radiation acute effects have disappeared.
* Hemoglobin equal or greater than 9 g/L. (allowed transfusion prior to treatment to reach this hemoglobin level).
* Leukocytes greater or equal to 4000/mm3.
* Platelets equal or greater to 100 000 mm3.
* Hepatic: Total bilirubin up to 1.5 times normal value, albumin equal or greater to 2: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) lower or equal to 2.5 times the regular superior limit.
* Renal: Normal creatinine. If high, the extent debugging must be greater than 60 mL/min.
* With the exception of alopecia, patients should have resolution of all acute toxic effects of any prior surgery, radiotherapy or chemotherapy, such effects qualified according to the Common Toxicity Criteria (CTC version 3.0) from the National Cancer Institute (NCI), or within the limits shown in laboratory parameters mentioned above.
* Be willing and able to comply with the programmed visits, the treatment plan and laboratory tests.
* The ability to understand the nature of the study and give a report written consent.

Exclusion Criteria:

* Small cell and/or neuroendocrine cervical cancer.
* History of allergy to hydralazine, magnesium valproate or sulfa.
* Any disease of collagen present (Systemic Lupus Erythematosus (SLE), Rheumatoid arthritis (RA), etc), or history of the same.
* Recent or past condition of symptomatic postural hypotension diagnosed by a clinician.
* Secondary heart failure to aortic stenosis or any other condition where a vasodilator is contraindicated.
* Recent or past condition of active disease of the central nervous system, including seizures.
* Previous or current use of magnesium valproate and/or any other anticonvulsive.
* Pregnant patients or nursing.
* Prior cancer within the last 5 years or in presence of a second primary tumor (except carcinoma of the cervix in situ or basal cell carcinoma of the skin adequately treated).
* Use of any of the research agents in the month prior to enrollment in this study.
* Serious concomitant systemic disorders incompatible with the study at the discretion of the investigator.
* Recently receiving another onco-specific treatment research.
* The recently or previously diagnosed hypertension and controlled with any antihypertensive or a combination of them (provided that they do not include hydralazine) WON'T be an exclusion criteria.

Criteria Treatment Interruption

* A patient will be discontinued from the study under the following circumstances.
* If there is evidence of disease progression.
* Unacceptable toxicity.
* If the clinician considers that a change of therapy will be for the best interest of the patient.
* If the patient requests the discontinuation.
* If a patient gets pregnant or does not use an adequate birth control (for patients able to conceive).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  patient´s survival since inclusion in the study until final event of death.

SECONDARY OUTCOMES:
Objective Response | 6 months
  The treatment response will be evaluated according to the new international criteria from response evaluation committee in solid tumors (RECIST) (EJC 2009; 45:228-247). Objective Response will be evaluated after cycles 3 and 6 and every 3 months the first 2 years, every 4 months the third year, every 6 months the fourth year and later annually or until progression.
Toxicity | 7 months
  Haematological toxicity will be evaluated every 3 weeks during QT and every 3 months at Follow up according Common Terminology Criteria for Adverse Events (CTCAE) V.3.0 spanish.
Quality of life | 24 months
  Quality of life will be evaluated according the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire QLQ-C30 and QLQ-Cx24. Quality of life will be evaluated after cycles 3 and 6 of chemotherapy and every 6 months at follow up.
Progression free survival | 24 months
  Time after treatment in wich disease remains unprogressive. Progression free survival will be evaluated through objective response after cycles 3 and 6 and every 3 months every 3 months the first 2 years, every 4 months the third year, every 6 months the fourth year and later annually or until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Cetina Lucely, MSc, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- National Institute of Cancerology, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Bruner DW, Wasserman T. The impact on quality of life by radiation late effects. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1353-5. doi: 10.1016/0360-3016(95)00042-W. PMID 7713794
- [Background] Aaronson SA. Growth factors and cancer. Science. 1991 Nov 22;254(5035):1146-53. doi: 10.1126/science.1659742.
- [Background] Almonte M, Albero G, Molano M, Carcamo C, Garcia PJ, Perez G. Risk factors for human papillomavirus exposure and co-factors for cervical cancer in Latin America and the Caribbean. Vaccine. 2008 Aug 19;26 Suppl 11:L16-36. doi: 10.1016/j.vaccine.2008.06.008. PMID 18945400
- [Background] Arbyn M, Castellsague X, de Sanjose S, Bruni L, Saraiya M, Bray F, Ferlay J. Worldwide burden of cervical cancer in 2008. Ann Oncol. 2011 Dec;22(12):2675-2686. doi: 10.1093/annonc/mdr015. Epub 2011 Apr 6. PMID 21471563
- [Background] Arce C, Perez-Plasencia C, Gonzalez-Fierro A, de la Cruz-Hernandez E, Revilla-Vazquez A, Chavez-Blanco A, Trejo-Becerril C, Perez-Cardenas E, Taja-Chayeb L, Bargallo E, Villarreal P, Ramirez T, Vela T, Candelaria M, Camargo MF, Robles E, Duenas-Gonzalez A. A proof-of-principle study of epigenetic therapy added to neoadjuvant doxorubicin cyclophosphamide for locally advanced breast cancer. PLoS One. 2006 Dec 20;1(1):e98. doi: 10.1371/journal.pone.0000098. PMID 17183730
- [Background] Biancotto C, Frige G, Minucci S. Histone modification therapy of cancer. Adv Genet. 2010;70:341-86. doi: 10.1016/B978-0-12-380866-0.60013-7. PMID 20920755
- [Background] Candelaria M, Cetina L, Perez-Cardenas E, de la Cruz-Hernandez E, Gonzalez-Fierro A, Trejo-Becerril C, Taja-Chayeb L, Chanona J, Arias D, Duenas-Gonzalez A. Epigenetic therapy and cisplatin chemoradiation in FIGO stage IIIB cervical cancer. Eur J Gynaecol Oncol. 2010;31(4):386-91. PMID 20882878
- [Background] Candelaria M, Gallardo-Rincon D, Arce C, Cetina L, Aguilar-Ponce JL, Arrieta O, Gonzalez-Fierro A, Chavez-Blanco A, de la Cruz-Hernandez E, Camargo MF, Trejo-Becerril C, Perez-Cardenas E, Perez-Plasencia C, Taja-Chayeb L, Wegman-Ostrosky T, Revilla-Vazquez A, Duenas-Gonzalez A. A phase II study of epigenetic therapy with hydralazine and magnesium valproate to overcome chemotherapy resistance in refractory solid tumors. Ann Oncol. 2007 Sep;18(9):1529-38. doi: 10.1093/annonc/mdm204. PMID 17761710
- [Background] Candelaria M, Herrera A, Labardini J, Gonzalez-Fierro A, Trejo-Becerril C, Taja-Chayeb L, Perez-Cardenas E, de la Cruz-Hernandez E, Arias-Bofill D, Vidal S, Cervera E, Duenas-Gonzalez A. Hydralazine and magnesium valproate as epigenetic treatment for myelodysplastic syndrome. Preliminary results of a phase-II trial. Ann Hematol. 2011 Apr;90(4):379-87. doi: 10.1007/s00277-010-1090-2. Epub 2010 Oct 5. PMID 20922525
- [Background] Castellsague X, Munoz N. Chapter 3: Cofactors in human papillomavirus carcinogenesis--role of parity, oral contraceptives, and tobacco smoking. J Natl Cancer Inst Monogr. 2003;(31):20-8. PMID 12807941
- [Background] Chavez-Blanco A, Segura-Pacheco B, Perez-Cardenas E, Taja-Chayeb L, Cetina L, Candelaria M, Cantu D, Gonzalez-Fierro A, Garcia-Lopez P, Zambrano P, Perez-Plasencia C, Cabrera G, Trejo-Becerril C, Angeles E, Duenas-Gonzalez A. Histone acetylation and histone deacetylase activity of magnesium valproate in tumor and peripheral blood of patients with cervical cancer. A phase I study. Mol Cancer. 2005 Jul 7;4(1):22. doi: 10.1186/1476-4598-4-22. PMID 16001982
- [Background] Choi JI, Kim SH, Seong CK, Sim JS, Lee HJ, Do KH. Recurrent uterine cervical carcinoma: spectrum of imaging findings. Korean J Radiol. 2000 Oct-Dec;1(4):198-207. doi: 10.3348/kjr.2000.1.4.198. PMID 11752955
- [Background] Cull A, Cowie VJ, Farquharson DI, Livingstone JR, Smart GE, Elton RA. Early stage cervical cancer: psychosocial and sexual outcomes of treatment. Br J Cancer. 1993 Dec;68(6):1216-20. doi: 10.1038/bjc.1993.507. PMID 8260376
- [Background] de Villiers EM. Relationship between steroid hormone contraceptives and HPV, cervical intraepithelial neoplasia and cervical carcinoma. Int J Cancer. 2003 Mar 1;103(6):705-8. doi: 10.1002/ijc.10868. PMID 12516087
- [Background] Duenas-Gonzalez A, Candelaria M, Perez-Plascencia C, Perez-Cardenas E, de la Cruz-Hernandez E, Herrera LA. Valproic acid as epigenetic cancer drug: preclinical, clinical and transcriptional effects on solid tumors. Cancer Treat Rev. 2008 May;34(3):206-22. doi: 10.1016/j.ctrv.2007.11.003. Epub 2008 Jan 15. PMID 18226465
- [Background] Dueñas-Gonzalez A, Hinojosa García LM. Papel de la quimioterapia en el carcinoma cervicouterino. Rev Inst Nac Cancerol 46: 47-57, 2000.
- [Background] Duenas-Gonzalez A, Cetina L, Coronel J, Cervantes-Madrid D. Emerging drugs for cervical cancer. Expert Opin Emerg Drugs. 2012 Jun;17(2):203-18. doi: 10.1517/14728214.2012.683409. Epub 2012 Apr 25. PMID 22530838
- [Background] Duenas-Gonzalez A, Cetina L, Coronel J, Martinez-Banos D. Pharmacotherapy options for locally advanced and advanced cervical cancer. Drugs. 2010 Mar 5;70(4):403-32. doi: 10.2165/11534370-000000000-00000. PMID 20205484
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978
- [Background] Flores YN, Bishai DM, Shah KV, Lazcano-Ponce E, Lorincz A, Hernandez M, Ferris D, Salmeron J. Risk factors for cervical cancer among HPV positive women in Mexico. Salud Publica Mex. 2008 Jan-Feb;50(1):49-58. doi: 10.1590/s0036-36342008000100011. PMID 18297182
- [Background] Insinga RP, Perez G, Wheeler CM, Koutsky LA, Garland SM, Leodolter S, Joura EA, Ferris DG, Steben M, Hernandez-Avila M, Brown DR, Elbasha E, Munoz N, Paavonen J, Haupt RM; FUTURE I Investigators. Incident cervical HPV infections in young women: transition probabilities for CIN and infection clearance. Cancer Epidemiol Biomarkers Prev. 2011 Feb;20(2):287-96. doi: 10.1158/1055-9965.EPI-10-0791. PMID 21300618
- [Background] Friedlander M, Grogan M; U.S. Preventative Services Task Force. Guidelines for the treatment of recurrent and metastatic cervical cancer. Oncologist. 2002;7(4):342-7. PMID 12185296
- [Background] Goncalves A, Fabbro M, Lhomme C, Gladieff L, Extra JM, Floquet A, Chaigneau L, Carrasco AT, Viens P. A phase II trial to evaluate gefitinib as second- or third-line treatment in patients with recurring locoregionally advanced or metastatic cervical cancer. Gynecol Oncol. 2008 Jan;108(1):42-6. doi: 10.1016/j.ygyno.2007.07.057. Epub 2007 Nov 5. PMID 17980406
- [Background] Gonzalez-Fierro A, Vasquez-Bahena D, Taja-Chayeb L, Vidal S, Trejo-Becerril C, Perez-Cardenas E, de la Cruz-Hernandez E, Chavez-Blanco A, Gutierrez O, Rodriguez D, Fernandez Z, Duenas-Gonzalez A. Pharmacokinetics of hydralazine, an antihypertensive and DNA-demethylating agent, using controlled-release formulations designed for use in dosing schedules based on the acetylator phenotype. Int J Clin Pharmacol Ther. 2011 Aug;49(8):519-24. doi: 10.5414/cp201526. PMID 21781652
- [Background] Holzner B, Kemmler G, Sperner-Unterweger B, Kopp M, Dunser M, Margreiter R, Marschitz I, Nachbaur D, Fleischhacker WW, Greil R. Quality of life measurement in oncology--a matter of the assessment instrument? Eur J Cancer. 2001 Dec;37(18):2349-56. doi: 10.1016/s0959-8049(01)00307-0. PMID 11720827
- [Background] Jayasekara H, Rajapaksa LC, Greimel ER. The EORTC QLQ-CX24 cervical cancer-specific quality of life questionnaire: psychometric properties in a South Asian sample of cervical cancer patients. Psychooncology. 2008 Oct;17(10):1053-7. doi: 10.1002/pon.1310. PMID 18203241
- [Background] Jit M, Gay N, Soldan K, Hong Choi Y, Edmunds WJ. Estimating progression rates for human papillomavirus infection from epidemiological data. Med Decis Making. 2010 Jan-Feb;30(1):84-98. doi: 10.1177/0272989X09336140. Epub 2009 Jun 12. PMID 19525483
- [Background] Kitagawa R, Katsumata N, Ando M, Shimizu C, Fujiwara Y, Yoshikawa H, Satoh T, Nakanishi T, Ushijima K, Kamura T. A multi-institutional phase II trial of paclitaxel and carboplatin in the treatment of advanced or recurrent cervical cancer. Gynecol Oncol. 2012 May;125(2):307-11. doi: 10.1016/j.ygyno.2012.02.009. Epub 2012 Feb 12. PMID 22333993
- [Background] Klee M, Thranov I, Machin D. Life after radiotherapy: the psychological and social effects experienced by women treated for advanced stages of cervical cancer. Gynecol Oncol. 2000 Jan;76(1):5-13. doi: 10.1006/gyno.1999.5644. PMID 10620434
- [Background] Kurtz JE, Hardy-Bessard AC, Deslandres M, Lavau-Denes S, Largillier R, Roemer-Becuwe C, Weber B, Guillemet C, Paraiso D, Pujade-Lauraine E. Cetuximab, topotecan and cisplatin for the treatment of advanced cervical cancer: A phase II GINECO trial. Gynecol Oncol. 2009 Apr;113(1):16-20. doi: 10.1016/j.ygyno.2008.12.040. Epub 2009 Feb 15. PMID 19232434
- [Background] Lazcano-Ponce E, Herrero R, Munoz N, Cruz A, Shah KV, Alonso P, Hernandez P, Salmeron J, Hernandez M. Epidemiology of HPV infection among Mexican women with normal cervical cytology. Int J Cancer. 2001 Feb 1;91(3):412-20. doi: 10.1002/1097-0215(20010201)91:33.0.co;2-m. PMID 11169968
- [Background] Lee JS, Kim HS, Park JT, Lee MC, Park CS. Expression of vascular endothelial growth factor in the progression of cervical neoplasia and its relation to angiogenesis and p53 status. Anal Quant Cytol Histol. 2003 Dec;25(6):303-11. PMID 14714296
- [Background] Lee SL, Tameru AM. A Mathematical Model of Human Papillomavirus (HPV) in the United States and its Impact on Cervical Cancer. J Cancer. 2012;3:262-8. doi: 10.7150/jca.4161. Epub 2012 Jun 9. PMID 22773930
- [Background] Long HJ 3rd, Bundy BN, Grendys EC Jr, Benda JA, McMeekin DS, Sorosky J, Miller DS, Eaton LA, Fiorica JV; Gynecologic Oncology Group Study. Randomized phase III trial of cisplatin with or without topotecan in carcinoma of the uterine cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2005 Jul 20;23(21):4626-33. doi: 10.1200/JCO.2005.10.021. Epub 2005 May 23. PMID 15911865
- [Background] Louie KS, Castellsague X, de Sanjose S, Herrero R, Meijer CJ, Shah K, Munoz N, Bosch FX; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Smoking and passive smoking in cervical cancer risk: pooled analysis of couples from the IARC multicentric case-control studies. Cancer Epidemiol Biomarkers Prev. 2011 Jul;20(7):1379-90. doi: 10.1158/1055-9965.EPI-11-0284. Epub 2011 May 24. PMID 21610224
- [Background] Mani S, Herceg Z. DNA demethylating agents and epigenetic therapy of cancer. Adv Genet. 2010;70:327-40. doi: 10.1016/B978-0-12-380866-0.60012-5. PMID 20920754
- [Background] Mohar A, Frias-Mendivil M. Epidemiology of cervical cancer. Cancer Invest. 2000;18(6):584-90. doi: 10.3109/07357900009012198. No abstract available. PMID 10923107
- [Background] Monk BJ, Mas Lopez L, Zarba JJ, Oaknin A, Tarpin C, Termrungruanglert W, Alber JA, Ding J, Stutts MW, Pandite LN. Phase II, open-label study of pazopanib or lapatinib monotherapy compared with pazopanib plus lapatinib combination therapy in patients with advanced and recurrent cervical cancer. J Clin Oncol. 2010 Aug 1;28(22):3562-9. doi: 10.1200/JCO.2009.26.9571. Epub 2010 Jul 6. PMID 20606083
- [Background] Monk BJ, Sill MW, Burger RA, Gray HJ, Buekers TE, Roman LD. Phase II trial of bevacizumab in the treatment of persistent or recurrent squamous cell carcinoma of the cervix: a gynecologic oncology group study. J Clin Oncol. 2009 Mar 1;27(7):1069-74. doi: 10.1200/JCO.2008.18.9043. Epub 2009 Jan 12. PMID 19139430
- [Background] Monk BJ, Sill MW, McMeekin DS, Cohn DE, Ramondetta LM, Boardman CH, Benda J, Cella D. Phase III trial of four cisplatin-containing doublet combinations in stage IVB, recurrent, or persistent cervical carcinoma: a Gynecologic Oncology Group study. J Clin Oncol. 2009 Oct 1;27(28):4649-55. doi: 10.1200/JCO.2009.21.8909. Epub 2009 Aug 31. PMID 19720909
- [Background] Moore DH, Blessing JA, McQuellon RP, Thaler HT, Cella D, Benda J, Miller DS, Olt G, King S, Boggess JF, Rocereto TF. Phase III study of cisplatin with or without paclitaxel in stage IVB, recurrent, or persistent squamous cell carcinoma of the cervix: a gynecologic oncology group study. J Clin Oncol. 2004 Aug 1;22(15):3113-9. doi: 10.1200/JCO.2004.04.170. PMID 15284262
- [Background] Moore KN, Herzog TJ, Lewin S, Giuntoli RL, Armstrong DK, Rocconi RP, Spannuth WA, Gold MA. A comparison of cisplatin/paclitaxel and carboplatin/paclitaxel in stage IVB, recurrent or persistent cervical cancer. Gynecol Oncol. 2007 May;105(2):299-303. doi: 10.1016/j.ygyno.2006.12.031. Epub 2007 Feb 14. PMID 17303230
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Munoz N, Franceschi S, Bosetti C, Moreno V, Herrero R, Smith JS, Shah KV, Meijer CJ, Bosch FX; International Agency for Research on Cancer. Multicentric Cervical Cancer Study Group. Role of parity and human papillomavirus in cervical cancer: the IARC multicentric case-control study. Lancet. 2002 Mar 30;359(9312):1093-101. doi: 10.1016/S0140-6736(02)08151-5. PMID 11943256
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964
- [Background] Palacio-Mejia LS, Rangel-Gomez G, Hernandez-Avila M, Lazcano-Ponce E. Cervical cancer, a disease of poverty: mortality differences between urban and rural areas in Mexico. Salud Publica Mex. 2003;45 Suppl 3:S315-25. doi: 10.1590/s0036-36342003000900005. PMID 14746024
- [Background] Peiretti M, Zapardiel I, Zanagnolo V, Landoni F, Morrow CP, Maggioni A. Management of recurrent cervical cancer: a review of the literature. Surg Oncol. 2012 Jun;21(2):e59-66. doi: 10.1016/j.suronc.2011.12.008. Epub 2012 Jan 14. PMID 22244884
- [Background] Sanchez-Barriga JJ. [Mortality trends from cervical cancer in the seven socioeconomic regions and the thirty two federative entities of Mexico, 2000-2008]. Gac Med Mex. 2012 Jan-Feb;148(1):42-51. Spanish. PMID 22367308
- [Background] Pectasides D, Fountzilas G, Papaxoinis G, Pectasides E, Xiros N, Sykiotis C, Koumarianou A, Psyrri A, Panayiotides J, Economopoulos T. Carboplatin and paclitaxel in metastatic or recurrent cervical cancer. Int J Gynecol Cancer. 2009 May;19(4):777-81. doi: 10.1111/IGC.0b013e3181a40a8b. PMID 19509587
- [Background] Omura GA, Blessing JA, Vaccarello L, Berman ML, Clarke-Pearson DL, Mutch DG, Anderson B. Randomized trial of cisplatin versus cisplatin plus mitolactol versus cisplatin plus ifosfamide in advanced squamous carcinoma of the cervix: a Gynecologic Oncology Group study. J Clin Oncol. 1997 Jan;15(1):165-71. doi: 10.1200/JCO.1997.15.1.165. PMID 8996138
- [Background] Lewis MJ. Análisis de la situación del cáncer cervicouterino en América Latina y el Caribe. Washington, D.C. Organización Panamericana de la Salud / Organización Mundial de la Salud (OPS/OMS); 2004:40.
- [Background] Santin AD, Sill MW, McMeekin DS, Leitao MM Jr, Brown J, Sutton GP, Van Le L, Griffin P, Boardman CH. Phase II trial of cetuximab in the treatment of persistent or recurrent squamous or non-squamous cell carcinoma of the cervix: a Gynecologic Oncology Group study. Gynecol Oncol. 2011 Sep;122(3):495-500. doi: 10.1016/j.ygyno.2011.05.040. PMID 21684583
- [Background] Schilder RJ, Sill MW, Lee YC, Mannel R. A phase II trial of erlotinib in recurrent squamous cell carcinoma of the cervix: a Gynecologic Oncology Group Study. Int J Gynecol Cancer. 2009 Jul;19(5):929-33. doi: 10.1111/IGC.0b013e3181a83467. PMID 19574787
- [Background] Sit AS, Kelley JL, Gallion HH, Kunschner AJ, Edwards RP. Paclitaxel and carboplatin for recurrent or persistent cancer of the cervix. Cancer Invest. 2004;22(3):368-73. doi: 10.1081/cnv-200029062. PMID 15493357
- [Background] Smith JS, Green J, Berrington de Gonzalez A, Appleby P, Peto J, Plummer M, Franceschi S, Beral V. Cervical cancer and use of hormonal contraceptives: a systematic review. Lancet. 2003 Apr 5;361(9364):1159-67. doi: 10.1016/s0140-6736(03)12949-2. PMID 12686037
- [Background] Tewari KS, Sill MW, Long HJ 3rd, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, Monk BJ. Improved survival with bevacizumab in advanced cervical cancer. N Engl J Med. 2014 Feb 20;370(8):734-43. doi: 10.1056/NEJMoa1309748. PMID 24552320
- [Background] Tinker AV, Bhagat K, Swenerton KD, Hoskins PJ. Carboplatin and paclitaxel for advanced and recurrent cervical carcinoma: the British Columbia Cancer Agency experience. Gynecol Oncol. 2005 Jul;98(1):54-8. doi: 10.1016/j.ygyno.2005.03.037. PMID 15904950
- [Background] Vaccarella S, Herrero R, Dai M, Snijders PJ, Meijer CJ, Thomas JO, Hoang Anh PT, Ferreccio C, Matos E, Posso H, de Sanjose S, Shin HR, Sukvirach S, Lazcano-Ponce E, Ronco G, Rajkumar R, Qiao YL, Munoz N, Franceschi S. Reproductive factors, oral contraceptive use, and human papillomavirus infection: pooled analysis of the IARC HPV prevalence surveys. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2148-53. doi: 10.1158/1055-9965.EPI-06-0556. PMID 17119039
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] Wright JD, Viviano D, Powell MA, Gibb RK, Mutch DG, Grigsby PW, Rader JS. Bevacizumab combination therapy in heavily pretreated, recurrent cervical cancer. Gynecol Oncol. 2006 Nov;103(2):489-93. doi: 10.1016/j.ygyno.2006.03.023. Epub 2006 May 2. PMID 16647106
- [Background] Zagouri F, Sergentanis TN, Chrysikos D, Filipits M, Bartsch R. Molecularly targeted therapies in cervical cancer. A systematic review. Gynecol Oncol. 2012 Aug;126(2):291-303. doi: 10.1016/j.ygyno.2012.04.007. Epub 2012 Apr 11. PMID 22504292
- [Background] Zambrano P, Segura-Pacheco B, Perez-Cardenas E, Cetina L, Revilla-Vazquez A, Taja-Chayeb L, Chavez-Blanco A, Angeles E, Cabrera G, Sandoval K, Trejo-Becerril C, Chanona-Vilchis J, Duenas-Gonzalez A. A phase I study of hydralazine to demethylate and reactivate the expression of tumor suppressor genes. BMC Cancer. 2005 Apr 29;5:44. doi: 10.1186/1471-2407-5-44. PMID 15862127